CLINICAL TRIAL: NCT00450125
Title: Six-Minute Walk Test in the Evaluation of Patients at High Risk for Complications From Lung Resection
Brief Title: Six-Minute Walk Test in Patients at High Risk for Complications From Lung Resection
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2006-1061
Record Dates: First submitted 2007-03-19; First posted 2007-03-21 (Estimated); Last update posted 2019-05-15 (Actual); Status verified 2018-09

CONDITIONS: Lung Cancer
Keywords: Lung Cancer; Lung Resection; Exercise Stress Test; Six-Minute Walk Test
MeSH Terms: conditions — Lung Neoplasms | interventions — Exercise Test

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Six-Minute Walk Test: Two Six-minute walk tests where total distance walked measured. Tests performed within 15 days of an exercise stress test.
  Interventions: Other: Six-Minute Walk Test; Other: Exercise stress test

INTERVENTIONS:
Other: Six-Minute Walk Test — Six-Minute walk tests at least one hour after vigorous exertion (such as exercise stress test) and at least 20 minutes in between the first and second six-minute walk tests
Other: Exercise stress test — Scheduled gold standard exercise test, i.e. stress test, cycle ergometry with incremental workloads or oxygen consumption exercise studies
  Other Names: Stress test; oxygen consumption exercise test; gold standard exercise test

SUMMARY:
The goal of this clinical research study is to compare the 6-minute walk test with the exercise stress test, in patients who may have lung surgery. Researchers want to find out if the 6-minute walk test is as good as the exercise stress test at predicting possible complications that may occur after lung surgery.

DETAILED DESCRIPTION:
Description of the Study Tests:

The exercise stress test is commonly used for predicting possible complications that may occur after lung surgery. The 6-minute walk test is a simpler test that does not require as much equipment.

6-Minute Walk Test: If you agree to take part in this research study, you will be asked to perform two 6-minute walk tests along with your routine exercise stress test. Both 6-minute walk tests will be done within 15 Days of the already scheduled exercise stress test if your clinical condition does not change during that time period. The 6-minute walk tests should be done at least 2 hours before or 1 hour after the exercise stress test. The second 6-minute walk test may be done 20 minutes after the first one. If you had a 6-minute walk test done within 15 Days before enrolling in the study, it can be used for the study.

To perform the 6-minute walk tests, you will walk as far as possible around cones on a flat indoor course that is about 40 yards long. You will walk at your own pace and can take breaks at any time if necessary. After the 6 minutes, the study staff will tell you the total distance you have walked.

Researchers will compare the distances you walked for the two 6-minute walk tests with the results of the exercise stress test. The walk test results will not affect your treatment plan.

Other Study Procedures:

Before and after the walk tests, the following procedures will be performed. Your blood pressure will be measured. You will be asked about any shortness of breath and/or fatigue you may have.

Before, during, and for about 1 minute after the walk tests, your heart rate will be measured. A device that looks like a clothespin will be placed on your finger to wear during this time, and it will measure the amount of oxygen in your blood.

Length of Study:

You will be considered off-study after the second walk test.

If you do have lung surgery, researchers will monitor your health status by checking your medical records until you are discharged from the hospital or for 30 days after the lung surgery, whichever comes first.

This is an investigational study. Using the 6-minute walk test for this study's purpose is considered experimental. Up to 101 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patient's age is between 18-90.
2. Patient has been referred for an oxygen consumption exercise test because they are considered high risk for morbidity and/or mortality post lung resection
3. Patient must be able to read, understand and provide informed consent.

Exclusion Criteria:

1. Patients diagnosed with angina pectoris
2. Patients diagnosed with critical aortic stenosis
3. Patients with unstable gait that persists with use of assistive device
4. Patients unable to walk

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients at high risk for complications from lung resection.
Sampling Method: Non-Probability Sample
Enrollment: 101 (Estimated)
Dates: Start 2007-02 (Actual); Primary Completion 2020-06-30 (Estimated); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
Correlation of pre-operative six-minute walk test results with that of the gold standard exercise test | Up to 15 days to complete 3 tests (two six-minute walk tests and a stress test)
  Results used to correlate the pre-operative six-minute walk test results with that of the gold standard exercise test (stress test) through analysis of gas exchange and measurement of oxygen uptake [oxygen volume (VO2)]. For the six-minute walk tests, recorded parameters are distance walked and pulse oximetry saturation percentage levels, and for gold standard exercise test, recorded are the gas exchange and measurement of oxygen uptake (VO2, ml/kg/min). Equivalence test performed to establish that the new test (six-minute walk) is comparable to the gold standard test (the VO2 peak) with an acceptable decreased sensitivity.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos A. Jimenez, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org